CLINICAL TRIAL: NCT07036939
Title: Efficacy and Safety of Bilateral Cervical Lymphatic-Venous Anastomosis in the Treatment of Multiple System Atrophy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Shengdi Chen, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-264
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Multiple System Atrophy
Keywords: Multiple system atrophy; glymphatic system; lymphatic-venous anastomosis
MeSH Terms: conditions — Multiple System Atrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate LVA group (Experimental): Participants will undergo bilateral cervical lymphatic-venous anastomosis (LVA) surgery within 2 weeks after baseline assessments (including clinical scales, biomarker testing, and neuroimaging).
  Interventions: Procedure: Immediate LVA
- Delayed LVA Group (Active Comparator): Identical LVA procedure performed at 6 months (±2 weeks) post-baseline
  Interventions: Procedure: Delayed LVA

INTERVENTIONS:
Procedure: Immediate LVA — Bilateral cervical lymphatic-venous anastomosis (LVA) performed within 2 weeks after baseline assessments.
  Arms: Immediate LVA group
Procedure: Delayed LVA — Identical LVA procedure performed at 6 months (±2 weeks) post-baseline
  Arms: Delayed LVA Group

SUMMARY:
Multiple System Atrophy (MSA) is a rare and aggressive neurodegenerative disorder characterized by a combination of motor impairments, autonomic dysfunction, and cerebellar ataxia, with no currently available disease-modifying therapies. Emerging evidence suggests that impaired glymphatic clearance of pathological α-synuclein aggregates may contribute to disease progression. This clinical study investigates the potential of bilateral cervical lymphatic-venous anastomosis (LVA) - a microsurgical procedure connecting deep cervical lymphatics to veins - to enhance glymphatic drainage and slow disease progression in MSA patients.

This single-center prospective clinical study will enroll patients with clinically confirmed MSA to undergo bilateral cervical lymphatic-venous anastomosis (LVA). Through comprehensive pre- and postoperative evaluations including clinical scale assessments, blood biomarker testing, and neuroimaging examinations, the study aims to evaluate the short-term and long-term effects of bilateral LVA on patients' motor function, autonomic symptoms, and quality of life, as well as its potential to delay disease progression.

The study will further investigate whether the potential clinical improvements from LVA are mediated through enhanced intracranial lymphatic drainage function and subsequent clearance of pathological α-Syn protein in the brain. Safety assessments will include monitoring and recording both short-term and long-term postoperative complications. This research may provide a novel non-pharmacological intervention approach for MSA treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meets the 2022 Chinese Expert Consensus Diagnostic Criteria for Clinically Established Multiple System Atrophy (MSA).
* Unified MSA Rating Scale Part IV (UMSARS-IV) global disability score ≤3.
* Age: 40-70 years
* ASA (American Society of Anesthesiologists) Physical Status Classification ≤III, indicating acceptable anesthesia risk.
* Ability to complete neuropsychological assessments, physical examinations, brain MRI, and venous blood sampling.
* Willing to participate, provide biospecimens, and sign informed consent.

Exclusion Criteria:

* Cognitive/Psychiatric Disorders: Congenital intellectual disability or severe neurological/psychiatric disorders affecting compliance.
* Severe Comorbidities: End-stage cardiac, hepatic, renal, or respiratory failure, or active malignancy with life expectancy <1 year.
* Surgical Contraindications:
* Coagulopathy (uncontrolled bleeding risk)
* Allergy to surgical drugs/contrast agents
* Active neck infection (skin/deep tissue)
* Inability to adhere to study visits.
* Participation in other competing clinical trials.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Bilateral LVA on MSA Symptoms at 3 Months (UMSARS-II Score Change) | Baseline to 3 months post-operation.
  Description:
  Change in Unified Multiple System Atrophy Rating Scale Part II (UMSARS-II) scores from baseline to 3 months post-LVA surgery.
  Scale Range: 0-56 (higher scores = worse motor function). Metric: Mean difference in total score.
Safety of Bilateral LVA (Surgical Adverse Events) | Intraoperative to 3 months post-operation.
  Incidence of surgery-related adverse events (e.g., infection, bleeding, anastomosis failure) within 3 months post-operation.
  Metric: Percentage of participants with ≥1 adverse event (AE).

SECONDARY OUTCOMES:
Long-term Efficacy of LVA on MSA Symptoms | Baseline to 6, 9, and 12 months post-operation.
  Change in UMSARS-II scores from baseline to 6, 9, and 12 months post-LVA. Scale Range: 0-56 (higher = worse). Metric: Mean difference at each timepoint.
Effect of LVA on Plasma Biomarkers | Baseline to 3 months post-operation.
  Change in plasma biomarkers from baseline to 3 months post-LVA. Metric: Concentration (pg/mL) via ELISA.
Assessment of Glymphatic Function via MRI ALPS Index | Preoperatively (baseline)，3 months post-LVA，12 months post-LVA
  Assessment of Glymphatic Function via MRI ALPS Index Glymphatic activity will be quantitatively evaluated using Diffusion Tensor Imaging along the Perivascular Space (DTI-ALPS) sequence on 3T MRI. The ALPS index will be calculated from diffusivity ratios (Dx/Dz) in the perivascular spaces of deep white matter (centrum semiovale level), reflecting interstitial fluid clearance efficiency. Higher ALPS indices indicate enhanced glymphatic function.
Cognitive Improvement Post-LVA | Baseline to 3, 6, 9, and 12 months post-operation.
  Change in Montreal Cognitive Assessment (MoCA) scores from baseline to 3/6/9/12 months.
  Scale Range: 0-30 (higher = better cognition).
Quality of Life Improvement | Baseline to 3, 6, 9, and 12 months post-operation.
  Change in Parkinson's Disease Questionnaire-39 (PDQ-39) scores from baseline to 3/6/9/12 months.
  Scale Range: 0-100 (lower = better QoL).
Disease-Modifying Effect of LVA (Delayed vs. Immediate Surgery) | Baseline， 3 Months，6 Months，9Months，and 12 Months
  Differences in Unified Multiple System Atrophy Rating Scale Part II (UMSARS-II) Changes from Baseline to 3 Months，6 Months，9Months，and 12 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided